CLINICAL TRIAL: NCT00002840
Title: PHASE III STUDY OF ADJUVANT PROCARBAZINE, CCNU AND VINCRISTINE CHEMOTHERAPY IN PATIENTS WITH HIGHLY ANAPLASTIC OLIGODENDROGLIOMA
Brief Title: Radiation Therapy With and Without Combination Chemotherapy in Patients With Resected Anaplastic Oligodendroglioma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-26951; EORTC-26951; MRC-BR11
Record Dates: First submitted 1999-11-01; First posted 2004-01-22 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult anaplastic oligodendroglioma; adult mixed glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Oligodendroglioma; Glioma | interventions — Lomustine; Procarbazine; Vincristine; Radiotherapy

INTERVENTIONS:
Drug: lomustine
Drug: procarbazine hydrochloride
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells, and may be an effective treatment for anaplastic oligodendroglioma. Combining combination chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare radiation therapy with and without combination chemotherapy in patients with resected anaplastic oligodendroglioma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare survival and time to first progression in patients with anaplastic oligodendroglioma treated with radiotherapy with or without adjuvant procarbazine, lomustine, and vincristine (PCV) following surgical resection. II. Investigate the effect of PCV on quality of life and neurologic function in these patients. III. Determine the toxicity of PCV in these patients. IV. Correlate chromosomal lesions (1p and/or 19q, 9p, p53 loss and mutation, amplification of chromosome 7, or loss of chromosome 10) with progression-free and overall survival in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age, extent of resection, performance status, prior surgery, and participating center. Patients are randomized to one of two treatment arms. Arm I: Within 4-6 weeks after surgery, patients undergo radiotherapy over 7 weeks to the residual tumor volume. Arm II: Patients undergo radiotherapy as in arm I, then begin chemotherapy within 4 weeks after the completion of radiotherapy. Patients receive oral lomustine on day 1, oral procarbazine on days 8-21, and vincristine IV on days 8 and 29. Treatment repeats every 6 weeks in stable and responding patients for a total of 6 courses. Patients with disease recurrence may receive 6 additional courses of chemotherapy as above or another modality at the investigator's discretion. Patients are followed every 3 months for 1 year and then every 6 months for survival.

PROJECTED ACCRUAL: A total of 350 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Newly diagnosed oligodendroglioma or oligoastrocytoma (with at least 25% oligodendral elements) Low-grade oligodendroastrocytoma or oligodendroglioma that is recurrent after surgery without radiotherapy is allowed Prior partial or gross total resection of tumor (or biopsy only in case of no further surgical option) required At least 3 of the following histologic anaplastic features: High cellularity Endothelial abnormalities Nuclear abnormalities Necrosis Mitoses

PATIENT CHARACTERISTICS: Age: 16 to 69 Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.4 mg/dL Renal: Creatinine no greater than 1.3 mg/dL Creatinine clearance at least 60 mL/min Other: Not pregnant or nursing Fertile patients must use effective contraception No active or uncontrolled infection No other disease, including malignancy, that would preclude study No neurologic or psychiatric disturbance that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics No prior radiotherapy to the skull Surgery: See Disease Characteristics

Ages: 16 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 1996-08; Primary Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin J. van Den Bent, MD, Study Chair — Daniel Den Hoed Cancer Center at Erasmus Medical Center
Locations (40):
- Kaiser Franz Josef Hospital, Vienna (Wien), Austria
- Belgium (4):
  - Hopital Universitaire Erasme, Brussels
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels (Bruxelles)
  - Hopital de Jolimont, Haine-Saint-Paul
  - U.Z. Gasthuisberg, Leuven
- Turku University Central Hospital, Turku, Finland
- France (10):
  - Centre Hospitalier Regional de Lille, Lille
  - CHU de la Timone, Marseille
  - CHU de Nancy - Hopital Neurologique, Nancy
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Hopital Pasteur, Nice
  - Centre Antoine Lacassagne, Nice
  - C.H.R. de Nimes - Hopital Caremeau, Nîmes
  - CHU Pitie-Salpetriere, Paris
  - Centre Eugene Marquis, Rennes
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Neurologische Klinik der Henriettenstiftung, Hanover
  - Klinikum der Friedrich-Schiller Universitaet Jena, Jena
- National Institute of Neurosurgery, Budapest, Hungary
- Italy (2):
  - Azienda Ospedaliera di Padova, Padova (Padua)
  - Universita di Padova, Padua
- Netherlands (9):
  - Medisch Centrum Haaglanden, 's-Gravenhage (Den Haag, the Hague)
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Academisch Ziekenhuis Groningen, Groningen
  - University Medical Center Nijmegen, Nijmegen
  - Rotterdam Cancer Institute, Rotterdam
  - St. Elisabeth Ziekenhuis, Tilburg
  - Dr. Bernard Verbeeten Instituut, Tilburg
  - Academisch Ziekenhuis Utrecht, Utrecht
- Instituto Portugues de Oncologia de Francisco Gentil, Lisbon, Portugal
- Sweden (2):
  - University Hospital of Linkoping, Linköping
  - Umea Universitet, Umeå
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- United Kingdom (6):
  - Nottingham General Hospital, Nottingham, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Queen's Medical Centre, Nottingham, England
  - Royal South Hants Hospital, Southampton, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden Hospital, Sutton, England

REFERENCES:
- [Result] Idbaih A, Dalmasso C, Kouwenhoven M, Jeuken J, Carpentier C, Gorlia T, Kros JM, French P, Teepen J, Broet P, Delattre O, Mokhtari K, Sanson M, Delattre JY, van den Bent M, Hoang-Xuan K. Genomic aberrations associated with outcome in anaplastic oligodendroglial tumors treated within the EORTC phase III trial 26951. J Neurooncol. 2011 Jun;103(2):221-30. doi: 10.1007/s11060-010-0380-9. Epub 2010 Sep 6. PMID 20820870
- [Result] Mokhtari K, Ducray F, Kros JM, Gorlia T, Idbaih A, Taphoorn M, Wesseling P, Hoang-Xuan K, Van den Bent M, Sanson M. Alpha-internexin expression predicts outcome in anaplastic oligodendroglial tumors and may positively impact the efficacy of chemotherapy: European organization for research and treatment of cancer trial 26951. Cancer. 2011 Jul 1;117(13):3014-26. doi: 10.1002/cncr.25827. Epub 2011 Jan 18. PMID 21246521
- [Result] van den Bent MJ, Gravendeel LA, Gorlia T, Kros JM, Lapre L, Wesseling P, Teepen JL, Idbaih A, Sanson M, Smitt PA, French PJ. A hypermethylated phenotype is a better predictor of survival than MGMT methylation in anaplastic oligodendroglial brain tumors: a report from EORTC study 26951. Clin Cancer Res. 2011 Nov 15;17(22):7148-55. doi: 10.1158/1078-0432.CCR-11-1274. Epub 2011 Sep 13. PMID 21914791
- [Result] Preusser M, Hoeftberger R, Woehrer A, et al.: Prognostic value and analytical performance (reproducibility) of Ki67 index in anaplastic oligodendroglial tumors: A translational study of the EORTC Brain Tumor Group. [Abstract] J Clin Oncol 28 (Suppl 15): A-2029, 2010.
- [Result] van den Bent MJ, Dubbink HJ, Marie Y, Brandes AA, Taphoorn MJ, Wesseling P, Frenay M, Tijssen CC, Lacombe D, Idbaih A, van Marion R, Kros JM, Dinjens WN, Gorlia T, Sanson M. IDH1 and IDH2 mutations are prognostic but not predictive for outcome in anaplastic oligodendroglial tumors: a report of the European Organization for Research and Treatment of Cancer Brain Tumor Group. Clin Cancer Res. 2010 Mar 1;16(5):1597-604. doi: 10.1158/1078-0432.CCR-09-2902. Epub 2010 Feb 16. PMID 20160062
- [Result] Kouwenhoven MC, Gorlia T, Kros JM, Ibdaih A, Brandes AA, Bromberg JE, Mokhtari K, van Duinen SG, Teepen JL, Wesseling P, Vandenbos F, Grisold W, Sipos L, Mirimanoff R, Vecht CJ, Allgeier A, Lacombe D, van den Bent MJ. Molecular analysis of anaplastic oligodendroglial tumors in a prospective randomized study: A report from EORTC study 26951. Neuro Oncol. 2009 Dec;11(6):737-46. doi: 10.1215/15228517-2009-011. PMID 19224764
- [Result] van den Bent MJ, Dubbink HJ, Sanson M, van der Lee-Haarloo CR, Hegi M, Jeuken JW, Ibdaih A, Brandes AA, Taphoorn MJ, Frenay M, Lacombe D, Gorlia T, Dinjens WN, Kros JM. MGMT promoter methylation is prognostic but not predictive for outcome to adjuvant PCV chemotherapy in anaplastic oligodendroglial tumors: a report from EORTC Brain Tumor Group Study 26951. J Clin Oncol. 2009 Dec 10;27(35):5881-6. doi: 10.1200/JCO.2009.24.1034. Epub 2009 Nov 9. PMID 19901104
- [Result] Kros JM, Gorlia T, Kouwenhoven MC, Zheng PP, Collins VP, Figarella-Branger D, Giangaspero F, Giannini C, Mokhtari K, Mork SJ, Paetau A, Reifenberger G, van den Bent MJ. Panel review of anaplastic oligodendroglioma from European Organization For Research and Treatment of Cancer Trial 26951: assessment of consensus in diagnosis, influence of 1p/19q loss, and correlations with outcome. J Neuropathol Exp Neurol. 2007 Jun;66(6):545-51. doi: 10.1097/01.jnen.0000263869.84188.72. PMID 17549014
- [Result] Mauer ME, Taphoorn MJ, Bottomley A, Coens C, Efficace F, Sanson M, Brandes AA, van der Rijt CC, Bernsen HJ, Frenay M, Tijssen CC, Lacombe D, van den Bent MJ; EORTC Brain Cancer Group. Prognostic value of health-related quality-of-life data in predicting survival in patients with anaplastic oligodendrogliomas, from a phase III EORTC brain cancer group study. J Clin Oncol. 2007 Dec 20;25(36):5731-7. doi: 10.1200/JCO.2007.11.1476. PMID 18089867
- [Result] Taphoorn MJ, van den Bent MJ, Mauer ME, Coens C, Delattre JY, Brandes AA, Sillevis Smitt PA, Bernsen HJ, Frenay M, Tijssen CC, Lacombe D, Allgeier A, Bottomley A; European Organisation for Research and Treatment of Cancer. Health-related quality of life in patients treated for anaplastic oligodendroglioma with adjuvant chemotherapy: results of a European Organisation for Research and Treatment of Cancer randomized clinical trial. J Clin Oncol. 2007 Dec 20;25(36):5723-30. doi: 10.1200/JCO.2007.12.7514. PMID 18089866
- [Result] van den Bent MJ, Carpentier AF, Brandes AA, Sanson M, Taphoorn MJ, Bernsen HJ, Frenay M, Tijssen CC, Grisold W, Sipos L, Haaxma-Reiche H, Kros JM, van Kouwenhoven MC, Vecht CJ, Allgeier A, Lacombe D, Gorlia T. Adjuvant procarbazine, lomustine, and vincristine improves progression-free survival but not overall survival in newly diagnosed anaplastic oligodendrogliomas and oligoastrocytomas: a randomized European Organisation for Research and Treatment of Cancer phase III trial. J Clin Oncol. 2006 Jun 20;24(18):2715-22. doi: 10.1200/JCO.2005.04.6078. PMID 16782911
- [Result] van den Bent MJ, Delattre JY, Brandes AA, et al.: First analysis of EORTC trial 26951, a randomized phase III study of adjuvant PCV chemotherapy in patients with highly anaplastic oligodendroglioma. [Abstract] J Clin Oncol 23 (Suppl 16): A-1503, 114s, 2005.
- [Derived] Lassman AB, Hoang-Xuan K, Polley MC, Brandes AA, Cairncross JG, Kros JM, Ashby LS, Taphoorn MJB, Souhami L, Dinjens WNM, Laack NN, Kouwenhoven MCM, Fink KL, French PJ, Macdonald DR, Lacombe D, Won M, Gorlia T, Mehta MP, van den Bent MJ. Joint Final Report of EORTC 26951 and RTOG 9402: Phase III Trials With Procarbazine, Lomustine, and Vincristine Chemotherapy for Anaplastic Oligodendroglial Tumors. J Clin Oncol. 2022 Aug 10;40(23):2539-2545. doi: 10.1200/JCO.21.02543. Epub 2022 Jun 22. PMID 35731991
- [Derived] Erdem-Eraslan L, Gravendeel LA, de Rooi J, Eilers PH, Idbaih A, Spliet WG, den Dunnen WF, Teepen JL, Wesseling P, Sillevis Smitt PA, Kros JM, Gorlia T, van den Bent MJ, French PJ. Intrinsic molecular subtypes of glioma are prognostic and predict benefit from adjuvant procarbazine, lomustine, and vincristine chemotherapy in combination with other prognostic factors in anaplastic oligodendroglial brain tumors: a report from EORTC study 26951. J Clin Oncol. 2013 Jan 20;31(3):328-36. doi: 10.1200/JCO.2012.44.1444. Epub 2012 Dec 26. PMID 23269986
- [Derived] van den Bent MJ, Brandes AA, Taphoorn MJ, Kros JM, Kouwenhoven MC, Delattre JY, Bernsen HJ, Frenay M, Tijssen CC, Grisold W, Sipos L, Enting RH, French PJ, Dinjens WN, Vecht CJ, Allgeier A, Lacombe D, Gorlia T, Hoang-Xuan K. Adjuvant procarbazine, lomustine, and vincristine chemotherapy in newly diagnosed anaplastic oligodendroglioma: long-term follow-up of EORTC brain tumor group study 26951. J Clin Oncol. 2013 Jan 20;31(3):344-50. doi: 10.1200/JCO.2012.43.2229. Epub 2012 Oct 15. PMID 23071237